CLINICAL TRIAL: NCT03375437
Title: RNASARC - Molecular Screening Program of Soft Tissue Sarcomas With Complex Genomic Profile to Detect NTRK1/2/3, ROS1 or ALK Gene Fusions.
Acronym: RNASARC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ET17-080 (RNASARC)
Record Dates: First submitted 2017-12-04; First posted 2017-12-18 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Soft Tissue Sarcoma; Advanced Cancer; Metastatic Cancer
Keywords: Clinical Trial; Multicenter Trial; NTRK1; NTRK2; NTRK3; ROS1; ALK; RNAseq; entrectinib; STARTRK-2
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NTRK, ROS and ALK molecular screening (Experimental): The molecular screening to detect NTRK1, 2, 3, ROS or ALK gene rearrangements will be a two step process, consisting of:
  1. First, immunohistochemistry (IHC) assay to detect protein expression of TRKA/B/C (encoded by NRTK1,2,3), ROS1 or ALK.
  2. Second, RNAseq analysis will be performed on positive IHC specimens to detect specific rearrangements in the NTRK1, NTRK2, NTRK3, ROS1 or ALK genes.
  Interventions: Genetic: Blood and tumor samples

INTERVENTIONS:
Genetic: Blood and tumor samples — FFPE tumor block (archival or a dedicated freshly collected tumor biopsy) will be collected for all enrolled patients and centralized.
  Blood sampling for Translational Research (optional) (2*10mL EDTA)

SUMMARY:
This trial is a multicenter, prospective cohort study aiming to describe molecular profiles of soft tissue sarcoma (STS) with complex genomic profiles in particular to assess the incidence of NTRK1/2/3, ROS1 or ALK gene fusions to direct such patients through an ongoing clinical trial with entrectinib when appropriate. An exploratory translational program is also correlated to this trial in order to analyse immune gene expression.

DETAILED DESCRIPTION:
Following inform consent form (ICF) signature, a formalin-fixed and paraffin-embedded (FFPE) tumor block (archival or a dedicated freshly collected tumor biopsy) will be collected for all enrolled patients and centralized at the biological resources platform of the Centre Léon Bérard.

At reception, a central pathological review will be performed to confirm if quality and quantity of material is acceptable: all tumor sample should present at least 20 % (ideally 30 %) of tumor cells and have a surface area > 5 mm2 (optimal condition is a surface area of 5-25 mm2). If the quality and quantity of tumor sample do not meet the standards, patients will be considered as "screening failure". If standards are met, inclusion will be confirmed and molecular screening will be initiated as well as the translational research program.

The molecular screening to detect NTRK1,2,3, ROS1 or ALK gene rearrangements will be a two-step process, consisting of :

1. First, immunohistochemistry (IHC) assay to detect protein expression of TRKA/B/C (encoded by NTRK1,2,3), ROS1 or ALK. Only positive IHC samples will continued the 2nd step of molecular screening. Negative IHC patients do not require further NTRK, ROS or ALK gene rearrangement testing; however tumor samples will be further used for additional translational research program presented in Section VII and data about the clinical evolution of these patients will be collected
2. Second, RNAseq analysis will be performed on positive IHC specimens to detect specific rearrangements in the NTRK1,NTRK2, NTRK3, ROS1 or ALK genes.
3. Following molecular analyses, screening results will be immediately (within 24 hours) communicated to investigators, GSF-GETO Network and Ignyta representatives in order to recommend patients with NTRK1, NTRK2, NTRK3, ROS1 or ALK rearrangement for formal eligibility determination for potential enrolment in a clinical trial in particular with entrectinib (STARTRK-2; NCT02568267).

ELIGIBILITY:
Inclusion Criteria:

* I1. Male or female patients aged ≥ 12 years at time of informed consent form (ICF) signature.
* I2. Histologically confirmed diagnosis of advanced /metastatic disease STS with complex genomics (e.g., Leiomyosarcoma [LMS], Undifferentiated Pleomorphic Sarcoma [UPS], pleomorphic liposarcoma/rhabdomyosarcoma [P-LPS/P-RMS], angiosarcoma, malignant peripheral nerve sheath tumor [MPNST], myxofibrosarcoma, fibrosarcoma).
* I3. Availability of a representative formalin-fixed, paraffin-embedded (FFPE) tumor sample, with the corresponding hematoxylin and eosin stained slide and a pathological report:

either a tumor archival block (less than 3 years old) or a dedicated freshly collected de novo biopsy performed from one accessible lesion visible by medical imaging and accessible to percutaneous sampling with a diameter of at least 10 mm.

* I4. Tumor sample meeting following quality/quantity control (QC) criteria confirmed by a central pathological review:

at least 20% (ideally 30%) of tumor cells and a sample size surface area > 5mm2 (ideally 5-25mm2).

* I5. Patient (and legal guardians if not-emancipated minor) should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study procedures as per protocol.
* I6. Patient must be covered by a medical insurance.

Non-inclusion criteria:

* NI1. Patients with non-assessable tumor sample.
* NI2. Prior treatment with approved or investigational TRK, ROS1, or ALK inhibitors. Any other prior anticancer therapy are allowed with no limit of prior number of treatment lines.
* NI3. Pregnant or breast-feeding patients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with NTRK1/2/3, ROS1 or ALK gene fusions (95% confidence interval) | 24 months
  Such molecular pre-screening will allow to direct eligible patients with sarcomas harboring an NTRK1/2/3, ROS1 or ALK fusion to a clinical trial with entrectinib, when judged appropriate by the patient's treating oncologist. Depending of the molecular alterations, other therapeutic options could be envisaged.

SECONDARY OUTCOMES:
Proportion of patients with NTRK1/2/3, ROS1, or ALK gene fusion per histological sub-types of STS with complex genomics | 24 months since first inclusion
  the partitioning of STS patients with NTRK1/2/3, ROS1 or ALK gene fusions within the different STS sub-types.
Clinical characteristics of patients with NTRK1/2/3, ROS1, or ALK gene fusion versus patients with no NTRK1/2/3, ROS1, or ALK gene fusion. | 24 months since first inclusion
  Comparisons of quantitative variables will be assessed with Student t-test or Wilcoxon-Mann and Whitney test , as appropriate. Comparisons of qualitative variables will be assessed with the X2 test or the Fisher's exact test, as appropriate.
anti-cancer treatments initiated since inclusion. | 36 months
  anti-cancer treatments initiated since inclusion among patients with NTRK1/2/3, ROS1, or ALK gene fusion and among patients with no NTRK1/2/3, ROS1, or ALK gene fusion.
Overall survival (OS) | 36 months
  Overall survival (OS) among patients with NTRK1/2/3, ROS1, or ALK gene fusion and among patients with no NTRK1/2/3, ROS1, or ALK gene fusion. It will be measured from the date of STS diagnosis to the date of death from any cause. Patients who are alive at the time of analysis will be censored at the date of last contact. OS will be estimated using the Kaplan-Meier method, and will be described in terms of medians along with the associated 2-sided 95% confidence interval (CI)

CONTACTS AND LOCATIONS:
Overall Officials: Armelle DUFRESNE, MD, Principal Investigator — Centre Leon Berard
Locations (10):
- France (10):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHU de Limoges Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Lorraine, Nancy
  - Centre Antoine Lacassagne, Nice
  - Institut Gustave ROUSSY, Paris
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez

REFERENCES:
- [Background] Tap WD, Jones RL, Van Tine BA, Chmielowski B, Elias AD, Adkins D, Agulnik M, Cooney MM, Livingston MB, Pennock G, Hameed MR, Shah GD, Qin A, Shahir A, Cronier DM, Ilaria R Jr, Conti I, Cosaert J, Schwartz GK. Olaratumab and doxorubicin versus doxorubicin alone for treatment of soft-tissue sarcoma: an open-label phase 1b and randomised phase 2 trial. Lancet. 2016 Jul 30;388(10043):488-97. doi: 10.1016/S0140-6736(16)30587-6. Epub 2016 Jun 9. PMID 27291997
- [Background] Jain S, Xu R, Prieto VG, Lee P. Molecular classification of soft tissue sarcomas and its clinical applications. Int J Clin Exp Pathol. 2010 Apr 23;3(4):416-28. PMID 20490332
- [Background] Fleitas T, Ibarrola-Villava M, Ribas G, Cervantes A. MassARRAY determination of somatic oncogenic mutations in solid tumors: Moving forward to personalized medicine. Cancer Treat Rev. 2016 Sep;49:57-64. doi: 10.1016/j.ctrv.2016.07.007. Epub 2016 Jul 29. PMID 27501018
- [Background] Schmidt KT, Chau CH, Price DK, Figg WD. Precision Oncology Medicine: The Clinical Relevance of Patient-Specific Biomarkers Used to Optimize Cancer Treatment. J Clin Pharmacol. 2016 Dec;56(12):1484-1499. doi: 10.1002/jcph.765. Epub 2016 Jun 17. PMID 27197880
- [Background] Nakagawara A. Trk receptor tyrosine kinases: a bridge between cancer and neural development. Cancer Lett. 2001 Aug 28;169(2):107-14. doi: 10.1016/s0304-3835(01)00530-4. PMID 11431098
- [Background] Pulciani S, Santos E, Lauver AV, Long LK, Aaronson SA, Barbacid M. Oncogenes in solid human tumours. Nature. 1982 Dec 9;300(5892):539-42. doi: 10.1038/300539a0. No abstract available. PMID 7144906
- [Background] Martin-Zanca D, Hughes SH, Barbacid M. A human oncogene formed by the fusion of truncated tropomyosin and protein tyrosine kinase sequences. Nature. 1986 Feb 27-Mar 5;319(6056):743-8. doi: 10.1038/319743a0. PMID 2869410
- [Background] Shaw AT, Ou SH, Bang YJ, Camidge DR, Solomon BJ, Salgia R, Riely GJ, Varella-Garcia M, Shapiro GI, Costa DB, Doebele RC, Le LP, Zheng Z, Tan W, Stephenson P, Shreeve SM, Tye LM, Christensen JG, Wilner KD, Clark JW, Iafrate AJ. Crizotinib in ROS1-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Nov 20;371(21):1963-71. doi: 10.1056/NEJMoa1406766. Epub 2014 Sep 27. PMID 25264305
- [Background] Shaw AT, Kim DW, Mehra R, Tan DS, Felip E, Chow LQ, Camidge DR, Vansteenkiste J, Sharma S, De Pas T, Riely GJ, Solomon BJ, Wolf J, Thomas M, Schuler M, Liu G, Santoro A, Lau YY, Goldwasser M, Boral AL, Engelman JA. Ceritinib in ALK-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Mar 27;370(13):1189-97. doi: 10.1056/NEJMoa1311107. PMID 24670165
- [Background] Vaishnavi A, Le AT, Doebele RC. TRKing down an old oncogene in a new era of targeted therapy. Cancer Discov. 2015 Jan;5(1):25-34. doi: 10.1158/2159-8290.CD-14-0765. Epub 2014 Dec 19. PMID 25527197
- [Background] Doebele RC, Davis LE, Vaishnavi A, Le AT, Estrada-Bernal A, Keysar S, Jimeno A, Varella-Garcia M, Aisner DL, Li Y, Stephens PJ, Morosini D, Tuch BB, Fernandes M, Nanda N, Low JA. An Oncogenic NTRK Fusion in a Patient with Soft-Tissue Sarcoma with Response to the Tropomyosin-Related Kinase Inhibitor LOXO-101. Cancer Discov. 2015 Oct;5(10):1049-57. doi: 10.1158/2159-8290.CD-15-0443. Epub 2015 Jul 27. PMID 26216294
- [Result] Judson I, Verweij J, Gelderblom H, Hartmann JT, Schoffski P, Blay JY, Kerst JM, Sufliarsky J, Whelan J, Hohenberger P, Krarup-Hansen A, Alcindor T, Marreaud S, Litiere S, Hermans C, Fisher C, Hogendoorn PC, dei Tos AP, van der Graaf WT; European Organisation and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Doxorubicin alone versus intensified doxorubicin plus ifosfamide for first-line treatment of advanced or metastatic soft-tissue sarcoma: a randomised controlled phase 3 trial. Lancet Oncol. 2014 Apr;15(4):415-23. doi: 10.1016/S1470-2045(14)70063-4. Epub 2014 Mar 5. PMID 24618336
- [Result] Ryan CW, Merimsky O, Agulnik M, Blay JY, Schuetze SM, Van Tine BA, Jones RL, Elias AD, Choy E, Alcindor T, Keedy VL, Reed DR, Taub RN, Italiano A, Garcia Del Muro X, Judson IR, Buck JY, Lebel F, Lewis JJ, Maki RG, Schoffski P. PICASSO III: A Phase III, Placebo-Controlled Study of Doxorubicin With or Without Palifosfamide in Patients With Metastatic Soft Tissue Sarcoma. J Clin Oncol. 2016 Nov 10;34(32):3898-3905. doi: 10.1200/JCO.2016.67.6684. Epub 2016 Sep 30. PMID 27621408
- [Derived] Dufresne A, Pissaloux D, Ngo C, Penel N, Le Cesne A, Macagno N, Vanacker H, Henon C, Jean-Denis M, Rughoo K, Tirode F, Blay JY, Brahmi M. Natural history and treatment efficacy in an ambispective case series of NTRK-rearranged mesenchymal tumors. ESMO Open. 2023 Apr;8(2):101202. doi: 10.1016/j.esmoop.2023.101202. Epub 2023 Apr 11. PMID 37054503